CLINICAL TRIAL: NCT03570892
Title: Tisagenlecleucel Versus Standard of Care in Adult Patients With Relapsed or Refractory Aggressive B-cell Non-Hodgkin Lymphoma: A Randomized, Open Label, Phase III Trial (BELINDA)
Brief Title: Tisagenlecleucel in Adult Patients With Aggressive B-cell Non-Hodgkin Lymphoma
Acronym: BELINDA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CCTL019H2301; 2016-002966-29 (EudraCT Number); 2023-508343-48-00 (Registry Identifier: EU CTIS)
Record Dates: First submitted 2018-06-18; First posted 2018-06-27 (Actual); Results first posted 2024-07-23 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: Non-Hodgkin Lymphoma
Keywords: Non-Hodgkin's Lympoma; B-Cell Lymphoma; Diffuse Large B-cell Lymphoma; High Grade B-cell Lymphoma; Follicular Lymphoma grade 3B; CAR-T; Tisagenlecleucel; Kymriah; Immunotherapy; Cellular therapy; CTL019
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse | interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: Randomized, Open-Label
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tisagenlecleucel treatment strategy (Experimental): Patients received investigator's choice of optional platinum-based immunochemotherapy followed by lymphodepleting chemotherapy and a single dose of tisagenlecleucel
  Interventions: Drug: Tisagenlecleucel after optional bridging and lymphodepleting chemotherapy
- Standard of care treatment strategy (Active Comparator): Patients received investigator's choice of platinum-based immunochemotherapy followed in responding patients by high dose chemotherapy and autologous hematopoietic stem cell transplant (HSCT)
  Interventions: Drug: Platinum-based immunochemotherapy followed in responding patients with high dose chemotherapy and autologous hematopoietic stem cell transplant (HSCT)

INTERVENTIONS:
Drug: Tisagenlecleucel after optional bridging and lymphodepleting chemotherapy — Investigator's choice of optional platinum-based immunochemotherapy (ie. R-ICE, R-GemOx, R-GDP, R-DHAP) + Lymphodepleting chemotherapy (fludarabine with cyclophosphamide or bendamustine) + Tisagenlecleucel (a second generation CAR-T composed of a CD19 antigen-binding domain, a 4-1BB costimulatory domain and a CD3-ζ signaling domain)
  Arms: Tisagenlecleucel treatment strategy
Drug: Platinum-based immunochemotherapy followed in responding patients with high dose chemotherapy and autologous hematopoietic stem cell transplant (HSCT) — Investigator's choice of platinum-based immunochemotherapy (ie. R-ICE, R-GemOx, R-GDP, R-DHAP)+ High dose chemotherapy (ie. BEAM) + autologous HSCT.
  *Ibrutinib or lenalidomide may be used in patients who are no longer eligible for autologous HSCT after 2 cycles of immunochemotherapy
  Arms: Standard of care treatment strategy

SUMMARY:
This is a randomized, open label, multicenter phase III trial comparing the efficacy, safety, and tolerability of tisagenlecleucel to Standard Of Care in adult patients with aggressive B-cell Non-Hodgkin Lymphoma after failure of rituximab and anthracycline containing frontline immunochemotherapy.

DETAILED DESCRIPTION:
Approximately 318 subjects were planned to be randomized; 322 subjects were analyzed (Full analysis set): 162 subjects in the tisagenlecleucel arm and 160 subjects in the SOC arm.

The target population consisted of adult participants with aggressive B-cell non-Hodgkin lymphoma (NHL) who were relapsed/refractory within 365 days of their last dose of first line immunochemotherapy and eligible for autologous hematopoietic stem cell transplantation (HSCT).

The duration of treatment in the tisagenlecleucel treatment strategy is from the start of bridging chemotherapy (if applicable) until the infusion of tisagenlecleucel (expected on average at approximately 6 weeks from randomization). The duration of the treatment in the SOC treatment strategy is from the start of salvage chemotherapy until autologous HSCT. In either treatment arm, if infusion of tisagenlecleucel or autologous HSCT is not possible, the duration of treatment is until the last dose of study treatment prior to discontinuation of the treatment strategy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, aggressive B-cell NHL at relapse/progression or PR after front line therapy. Aggressive B-cell NHL is heretofore defined by the following list of subtypes (Swerdlow et al 2016):

  * DLBCL, NOS,
  * FL grade 3B,
  * Primary mediastinal large B cell lymphoma (PMBCL),
  * T cell rich/histiocyte rich large B cell lymphoma (T/HRBCL),
  * DLBCL associated with chronic inflammation,
  * Intravascular large B-cell lymphoma,
  * ALK+ large B-cell lymphoma,
  * B-cell lymphoma, unclassifiable, (with features intermediate between DLBCL and classical Hodgkin's Lymphoma (HL)),
  * High grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements,
  * High-grade B-cell lymphoma, NOS
  * HHV8+ DLBCL, NOS
  * DLBCL transforming from follicular lymphoma
  * DLBCL transforming from marginal zone lymphoma
  * DLBCL, leg type
* Relapse or progression within 365 days from last dose of anti CD20 antibody and anthracycline containing first line immunochemotherapy or refractory (have not achieved a CR).
* Patient is considered eligible for autologous HSCT as per local investigator assessment. Note: Intention to transplant and type of high dose chemotherapy (HDCT) regimen will be documented at the time of study entry
* Disease that is both active on PET scan (defined as 5-Deauville scorepoint-scale of 4 or 5) and measurable on CT scan, defined as::

  * Nodal lesions >15 mm in the long axis, regardless of the length of the short axis, and/or
  * Extranodal lesions (outside lymph node or nodal mass, but including liver and spleen) >10 mm in long AND short axis
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Adequate organ function:

Renal function defined as:

* Serum creatinine of ≤1.5 x upper limit of normal (ULN), OR estimated glomerular filtration rate (eGFR) ≥ 60 mL/min/1.73 m2

Hepatic function defined as:

* Alanine Transaminase (ALT) and Aspartate Transiminase (AST) ≤ 5 × ULN
* Total bilirubin ≤ 1.5 x ULN with the exception of patients with Gilbert syndrome who may be included if their total bilirubin is ≤3.0 × ULN and direct bilirubin ≤1.5 × ULN

Hematologic Function (regardless of transfusions) defined as:

* Absolute neutrophil count (ANC) >1000/mm3
* Absolute lymphocyte count (ALC) >300/mm3 OR Absolute number of CD3+ T cells >150/mm3 (only for patients with non-historical apheresis)
* Platelets ≥50000/mm3
* Hemoglobin >8.0 g/dl

Adequate pulmonary function defined as:

* No or mild dyspnea (≤ Grade 1)
* Oxygen saturation measured by pulse oximetry > 90% on room air
* Forced expiratory volume in 1 s (FEV1) ≥ 50% and/or carbon monoxide diffusion test (DLCO) ≥50% of predicted level - Must have a leukapheresis material of non-mobilized cells available for manufacturing.

Exclusion Criteria:

* Prior treatment with anti-CD19 therapy, T cell therapy, or any prior gene therapy product
* Treatment with any systemic lymphoma-directed second line anticancer therapy prior to randomization. Only steroids and local irradiation are permitted for disease control
* Patients with active central nervous system (CNS) involvement by disease under study are excluded, except if the CNS involvement has been effectively treated and local treatment was >4 weeks before randomization
* Prior allogeneic HSCT
* Clinically significant active infection
* Any of the following cardiovascular conditions:

  * Unstable angina, myocardial infarction, coronary artery bypass graft (CABG), or stroke within 6 months prior to screening,
  * Left ventricle ejection fraction (LVEF) <45% as determined by echocardiogram (ECHO) or magnetic resonance angiography (MRA) or multigated acquisition (MUGA) at the screening assessment.
  * New York Heart Association (NYHA) functional class III or IV (Chavey et al 2001), within the past 12 months.
  * Clinically significant cardiac arrhythmias (e.g., ventricular tachycardia), complete left bundle branch block, high-grade atrioventricular (AV) block (e.g., bifascicular block, Mobitz type II) and third degree AV block unless adequately controlled by pacemaker implantation.
  * Resting QTcF ≥450 msec (male) or ≥460 msec (female) at screening or inability to determine the QTcF interval
  * Risk factors for Torsades de Pointes (TdP), including uncorrected hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/ symptomatic bradycardia, or any of the following:
  * Long QT syndrome, family history of idiopathic sudden death or congenital long QT syndrome
  * Concomitant medication(s) with a "Known Risk of Torsades de Pointes" per crediblemeds.org that cannot be discontinued or replaced by safe alternative medication.
* Patients with active neurological autoimmune or inflammatory disorders (e.g., Guillain-Barré Syndrome (GBS), Amyotrophic Lateral Sclerosis (ALS)) and clinically significant active cerebrovascular disorders (e.g. cerebral edema, posterior reversible encephalopathy syndrome (PRES))

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2019-05-07 (Actual); Primary Completion 2021-05-06 (Actual); Study Completion 2026-02-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (69):
- United States (22):
  - Moores UC San Diego Cancer Center, La Jolla, California
  - University of California Los Angeles, Los Angeles, California
  - UCSF Medical Center, San Francisco, California
  - Sarah Cannon Research Institute, Denver, Colorado
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Booker Dynamic Brand Solutions, Atlanta, Georgia
  - Uni of Chi Medi Ctr Hema and Onco, Chicago, Illinois
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Wayne State University-Karmanos Cancer Institute, Detroit, Michigan
  - Uni of Nebraska Med Ctr, Omaha, Nebraska
  - Hackensack Uni Medical Center, Hackensack, New Jersey
  - Jewish Hospital, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
  - Oregon Health Sciences Univ, Portland, Oregon
  - Uni Pennsylvania Abramson Cncr Ctr, Philadelphia, Pennsylvania
  - MUSC Hollings Cancer Center, Charleston, South Carolina
  - Tennessee Oncology PLLC, Chattanooga, Tennessee
  - St Davids South Austin Medical Ctr, Austin, Texas
  - Texas Oncology-Baylor Scott and White, Dallas, Texas
  - Uni of Texas MD Anderson Ca Center, Houston, Texas
  - Methodist Hospital, San Antonio, Texas
  - Uni of Wisconsin Carbone Cancer Ctr, Madison, Wisconsin
- Australia (3):
  - Novartis Investigative Site, Darlinghurst, New South Wales
  - Novartis Investigative Site, Melbourne, Victoria
  - Novartis Investigative Site, Murdoch, Western Australia
- Austria (2):
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
- Novartis Investigative Site, Leuven, Belgium
- Brazil (2):
  - Novartis Investigative Site, Salvador, Estado de Bahia
  - Novartis Investigative Site, São Paulo
- China (2):
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
- France (6):
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pierre-Bénite
  - Novartis Investigative Site, Toulouse
- Germany (7):
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Leipzig, Saxony
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Ulm
- Novartis Investigative Site, Hong Kong, Hong Kong
- Italy (3):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Roma, RM
- Japan (6):
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Sendai, Miyagi
  - Tohoku University Hospital, Sendai, Miyagi
  - Novartis Investigative Site, Fukuoka
- Netherlands (4):
  - Novartis Investigative Site, Amsterdam, North Holland
  - Amsterdam UMC, locatie AMC, Amsterdam
  - Novartis Investigative Site, Utrecht
  - UMC Utrecht Cancer Center, Utrecht
- Novartis Investigative Site, Oslo, Norway
- Novartis Investigative Site, Singapore, Singapore
- Spain (4):
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Barcelona
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Salamanca
- Novartis Investigative Site, Zurich, Switzerland
- Novartis Investigative Site, Taipei, Taiwan
- United Kingdom (2):
  - Novartis Investigative Site, Birmingham, West Midlands
  - Novartis Investigative Site, London

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Bishop MR, Dickinson M, Purtill D, Barba P, Santoro A, Hamad N, Kato K, Sureda A, Greil R, Thieblemont C, Morschhauser F, Janz M, Flinn I, Rabitsch W, Kwong YL, Kersten MJ, Minnema MC, Holte H, Chan EHL, Martinez-Lopez J, Muller AMS, Maziarz RT, McGuirk JP, Bachy E, Le Gouill S, Dreyling M, Harigae H, Bond D, Andreadis C, McSweeney P, Kharfan-Dabaja M, Newsome S, Degtyarev E, Awasthi R, Del Corral C, Andreola G, Masood A, Schuster SJ, Jager U, Borchmann P, Westin JR. Second-Line Tisagenlecleucel or Standard Care in Aggressive B-Cell Lymphoma. N Engl J Med. 2022 Feb 17;386(7):629-639. doi: 10.1056/NEJMoa2116596. Epub 2021 Dec 14. PMID 34904798
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338
- [Derived] Thiruvengadam SK, Hunter B, Varnavski A, Fakhri B, Kaplan L, Ai WZ, Pampaloni M, Huang CY, Martin T 3rd, Damon L, Andreadis CB. Ofatumumab, Etoposide, and Cytarabine Intensive Mobilization Regimen in Patients with High-risk Relapsed/Refractory Diffuse Large B-Cell Lymphoma Undergoing Autologous Stem Cell Transplantation. Clin Lymphoma Myeloma Leuk. 2021 Apr;21(4):246-256.e2. doi: 10.1016/j.clml.2020.11.005. Epub 2020 Nov 11. PMID 33288485
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/34516954/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 18 countries and 65 sites. Approximately 318 subjects were planned to be randomized; 322 subjects were analyzed.
Pre-assignment Details: During the screening period, no lymphoma-specific therapy was allowed prior to randomization. During randomization, subjects were stratified by: Remission duration, international prognostic index (IPI) score and region.
Period: Overall Study
Arm/Group | Tisagenlecleucel Treatment Strategy | Standard of Care Treatment Strategy
Started | 162 | 160
Completed (Completed = Study on-going at the time of data cut-off date of 6-May-2021) | 105 | 106
Not Completed | 57 | 54
Not completed — Death | 51 | 45
Not completed — Subject decision | 5 | 3
Not completed — Protocol Violation | 1 | 4
Not completed — Physician Decision | 0 | 2

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) comprised all subjects to whom study treatment was assigned by randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tisagenlecleucel Treatment Strategy | Standard of Care Treatment Strategy | Total
Number analyzed (Participants) | 162 | 160 | 322
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (13.74) | 55.0 (12.99) | 55.8 (13.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 62 | 121
  Male | 103 | 98 | 201
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 128 | 128 | 256
  Asian | 20 | 22 | 42
  Black or African American | 8 | 3 | 11
  Unknown | 4 | 5 | 9
  American Indian or Alaska Native | 1 | 1 | 2
  Multiple | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival (EFS) Per Blinded Independent Review Committee (BIRC) Assessment
Description: Event-free survival (EFS) is defined as the time from the date of randomization to the date of the first documented disease progression or stable disease at or after the week 12 (+/- 1 week) assessment, as assessed by Blinded Independent Review Committee (BIRC) per Lugano criteria, or death due to any cause, at any time.
Time Frame: appro. 24 months
Population: The full analysis set (FAS) comprised all subjects to whom study treatment was assigned by randomization.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tisagenlecleucel Treatment Strategy | Standard of Care Treatment Strategy
Number analyzed (Participants) | 162 | 160
months | 3.0 [2.9 to 4.2] | 3.0 [3.0 to 3.5]
Statistical Analysis 1: Comparison: Tisagenlecleucel Treatment Strategy vs Standard of Care Treatment Strategy; Test type: Superiority; p = 0.694, Stratified log-rank test one-sided; Unadjusted stratified cox model hazard r = 1.07, 95% CI 2-sided [0.82 to 1.40]

2. Secondary Outcome: Event Free Survival (EFS) as Assessed by Local Investigator
Description: Event-free survival (EFS) is defined as the time from the date of randomization to the date of the first documented disease progression or stable disease.
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2027-02

3. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) is defined as the time from date of randomization to date of death due to any cause
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2027-02

4. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall Response Rate (ORR) as per the Lugano criteria as per BIRC review and local investigator assessment
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2027-02

5. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response: time from the date of first documented response of CR or PR to the date of first documented progression (SD or PD at or after the week 12 assessment will be considered progression) or death due to aggressive B-cell NHL. DOR will be summarized by BIRC and local response
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2027-02

6. Secondary Outcome: Time to Response (TTR)
Description: Time from the date of randomization to the date of a patient's first achieved a response of CR or PR on or after the Week 12 assessment
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2027-02

7. Secondary Outcome: SF-36v2
Description: Time to definitive deterioration in SF-36v2
Time Frame: 24 Months
Reporting Status: Not Posted, anticipated posting 2027-02

8. Secondary Outcome: FACT-Lym
Description: Time to definitive deterioration in FACT-Lym
Time Frame: 24 Months
Reporting Status: Not Posted, anticipated posting 2027-02

9. Secondary Outcome: EQ-VAS
Description: Time to definitive deterioration in EQ-VAS
Time Frame: 24 Months
Reporting Status: Not Posted, anticipated posting 2027-02

10. Secondary Outcome: Tisagenlecleucel Transgene Concentrations
Description: qPCR will be used to measure tisagenlecleucel transgene concentrations in peripheral blood and bone marrow
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2027-02

11. Secondary Outcome: Tisagenlecleucel Immunogenicity (Humoral and Cellular)
Description: Pre-existing and treatment related immunogenicity (humoral and cellular) of tisagenlecleucel will be characterized.
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2027-02

12. Secondary Outcome: Presence of Replication Competent Lentivirus (RCL)
Description: The presence of RCL will be assessed by VSV-qPCR in patients receiving tisagenlecleucel
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2027-02

ADVERSE EVENTS:
Time Frame: This primary analysis report includes data with a cut-off date 6-May-2021. Adverse Events (AEs) and death were collected from dose of study treatment to 56 days post last-infusion (defined as on-treatment) up to a max on-treatment period of approx. 2 years.
Description: Any sign or symptom that occurs during the conduct of the trial and safety follow-up.
  Other Adverse Event: An adverse event that is not a serious adverse event, meaning that it does not result in death, is not life-threatening, does not require inpatient hospitalization or extend a current hospital stay, does not result in an ongoing or significant incapacity or interfere substantially with normal life functions, and does not cause a congenital anomaly or birth defect.
Groups:
- All Participants: All participants who were enrolled in the study
Arm/Group | Tisagenlecleucel Treatment Strategy | Standard of Care Treatment Strategy | All Participants
All-Cause Mortality (participants affected / at risk) | 52/162 | 45/160 | 97/322
Serious Adverse Events (participants affected / at risk) | 76/162 | 82/160 | 158/322
Other Adverse Events (participants affected / at risk) | 159/162 | 158/160 | 317/322
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tisagenlecleucel Treatment Strategy (N=162) | Standard of Care Treatment Strategy (N=160) | All Participants (N=322)
Anaemia (Blood and lymphatic system disorders) | 2 | 7 | 9
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 0 | 1
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0 | 1
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 14 | 23 | 37
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 4 | 0 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2 | 3
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 2 | 4
Atrial flutter (Cardiac disorders) | 0 | 1 | 1
Cardiac arrest (Cardiac disorders) | 1 | 1 | 2
Mitral valve disease (Cardiac disorders) | 1 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 5 | 8
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0 | 2
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 | 1 | 1
Intestinal fistula (Gastrointestinal disorders) | 1 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 1
Mesenteric cyst (Gastrointestinal disorders) | 0 | 1 | 1
Nausea (Gastrointestinal disorders) | 3 | 4 | 7
Subileus (Gastrointestinal disorders) | 1 | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 3 | 5
Asthenia (General disorders) | 1 | 1 | 2
Catheter site inflammation (General disorders) | 0 | 1 | 1
Chest pain (General disorders) | 1 | 1 | 2
Disease progression (General disorders) | 6 | 2 | 8
Face oedema (General disorders) | 1 | 0 | 1
Fatigue (General disorders) | 2 | 0 | 2
Malaise (General disorders) | 0 | 1 | 1
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 1
Pain (General disorders) | 1 | 1 | 2
Pyrexia (General disorders) | 9 | 8 | 17
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 1
Hepatic failure (Hepatobiliary disorders) | 2 | 0 | 2
Anaphylactic shock (Immune system disorders) | 1 | 0 | 1
Cytokine release syndrome (Immune system disorders) | 22 | 0 | 22
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 | 0 | 1
Bacterial sepsis (Infections and infestations) | 3 | 0 | 3
COVID-19 (Infections and infestations) | 1 | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0 | 1
Device related infection (Infections and infestations) | 4 | 2 | 6
Enterococcal sepsis (Infections and infestations) | 1 | 0 | 1
Escherichia sepsis (Infections and infestations) | 1 | 0 | 1
Human herpesvirus 6 infection (Infections and infestations) | 0 | 1 | 1
Infection (Infections and infestations) | 0 | 1 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 2 | 3
Oral bacterial infection (Infections and infestations) | 1 | 0 | 1
Parainfluenzae virus infection (Infections and infestations) | 1 | 0 | 1
Pneumonia (Infections and infestations) | 3 | 1 | 4
Pneumonia cytomegaloviral (Infections and infestations) | 1 | 0 | 1
Pseudomonal sepsis (Infections and infestations) | 2 | 0 | 2
Sepsis (Infections and infestations) | 4 | 9 | 13
Septic shock (Infections and infestations) | 2 | 2 | 4
Staphylococcal sepsis (Infections and infestations) | 2 | 1 | 3
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 1 | 2
Urinary tract infection enterococcal (Infections and infestations) | 1 | 0 | 1
Acute haemolytic transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 0 | 2
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 | 1 | 1
Transfusion with incompatible blood (Injury, poisoning and procedural complications) | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1
Blood creatine increased (Investigations) | 1 | 0 | 1
Blood creatinine increased (Investigations) | 3 | 4 | 7
General physical condition abnormal (Investigations) | 1 | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0 | 1
Neutrophil count decreased (Investigations) | 2 | 2 | 4
Platelet count decreased (Investigations) | 2 | 5 | 7
White blood cell count decreased (Investigations) | 1 | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 2 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 3 | 4
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Central nervous system lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Sarcomatoid carcinoma of the lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1
Carotid artery stenosis (Nervous system disorders) | 1 | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 1 | 1
Hydrocephalus (Nervous system disorders) | 1 | 0 | 1
Immune effector cell-associated neurotoxicity syndrome (Nervous system disorders) | 1 | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 0 | 1 | 1
Myelitis transverse (Nervous system disorders) | 1 | 0 | 1
Neurotoxicity (Nervous system disorders) | 2 | 2 | 4
Paraplegia (Nervous system disorders) | 1 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 1
Spinal cord compression (Nervous system disorders) | 1 | 1 | 2
Syncope (Nervous system disorders) | 0 | 1 | 1
Bradyphrenia (Psychiatric disorders) | 1 | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 0 | 1
Substance-induced psychotic disorder (Psychiatric disorders) | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 3 | 6 | 9
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 1
Nephropathy toxic (Renal and urinary disorders) | 0 | 1 | 1
Prerenal failure (Renal and urinary disorders) | 0 | 1 | 1
Renal failure (Renal and urinary disorders) | 0 | 1 | 1
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Skin disorder (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 1
Hypertension (Vascular disorders) | 1 | 1 | 2
Hypotension (Vascular disorders) | 1 | 2 | 3
Hypovolaemic shock (Vascular disorders) | 0 | 1 | 1
Lymphatic fistula (Vascular disorders) | 0 | 1 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 1
Thrombophlebitis superficial (Vascular disorders) | 1 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1 | 1
Venous thrombosis (Vascular disorders) | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tisagenlecleucel Treatment Strategy (N=162) | Standard of Care Treatment Strategy (N=160) | All Participants (N=322)
Anaemia (Blood and lymphatic system disorders) | 80 | 114 | 194
Febrile neutropenia (Blood and lymphatic system disorders) | 9 | 22 | 31
Leukopenia (Blood and lymphatic system disorders) | 22 | 30 | 52
Lymphopenia (Blood and lymphatic system disorders) | 12 | 12 | 24
Neutropenia (Blood and lymphatic system disorders) | 67 | 65 | 132
Thrombocytopenia (Blood and lymphatic system disorders) | 59 | 78 | 137
Tachycardia (Cardiac disorders) | 11 | 3 | 14
Tinnitus (Ear and labyrinth disorders) | 2 | 9 | 11
Abdominal pain (Gastrointestinal disorders) | 15 | 25 | 40
Constipation (Gastrointestinal disorders) | 48 | 41 | 89
Diarrhoea (Gastrointestinal disorders) | 35 | 57 | 92
Nausea (Gastrointestinal disorders) | 67 | 78 | 145
Stomatitis (Gastrointestinal disorders) | 5 | 16 | 21
Vomiting (Gastrointestinal disorders) | 23 | 33 | 56
Asthenia (General disorders) | 8 | 18 | 26
Chills (General disorders) | 12 | 7 | 19
Fatigue (General disorders) | 38 | 49 | 87
Mucosal inflammation (General disorders) | 5 | 18 | 23
Oedema peripheral (General disorders) | 18 | 18 | 36
Pyrexia (General disorders) | 36 | 46 | 82
Cytokine release syndrome (Immune system disorders) | 78 | 0 | 78
Hypogammaglobulinaemia (Immune system disorders) | 16 | 7 | 23
Alanine aminotransferase increased (Investigations) | 10 | 11 | 21
Aspartate aminotransferase increased (Investigations) | 11 | 8 | 19
Blood alkaline phosphatase increased (Investigations) | 1 | 13 | 14
Blood creatinine increased (Investigations) | 28 | 28 | 56
C-reactive protein increased (Investigations) | 9 | 4 | 13
Lymphocyte count decreased (Investigations) | 6 | 9 | 15
Neutrophil count decreased (Investigations) | 40 | 28 | 68
Platelet count decreased (Investigations) | 36 | 50 | 86
White blood cell count decreased (Investigations) | 18 | 22 | 40
Decreased appetite (Metabolism and nutrition disorders) | 21 | 17 | 38
Hypocalcaemia (Metabolism and nutrition disorders) | 9 | 10 | 19
Hypokalaemia (Metabolism and nutrition disorders) | 45 | 48 | 93
Hypomagnesaemia (Metabolism and nutrition disorders) | 20 | 29 | 49
Hyponatraemia (Metabolism and nutrition disorders) | 12 | 9 | 21
Hypophosphataemia (Metabolism and nutrition disorders) | 13 | 17 | 30
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 9 | 22
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 10 | 25
Bone pain (Musculoskeletal and connective tissue disorders) | 9 | 14 | 23
Dizziness (Nervous system disorders) | 19 | 14 | 33
Headache (Nervous system disorders) | 37 | 31 | 68
Anxiety (Psychiatric disorders) | 10 | 9 | 19
Insomnia (Psychiatric disorders) | 15 | 12 | 27
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 12 | 29
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 20 | 33
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 10 | 13
Hiccups (Respiratory, thoracic and mediastinal disorders) | 7 | 12 | 19
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 | 8 | 21
Rash (Skin and subcutaneous tissue disorders) | 8 | 16 | 24
Hypertension (Vascular disorders) | 10 | 15 | 25
Hypotension (Vascular disorders) | 14 | 15 | 29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e., data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/92/NCT03570892/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-26): https://cdn.clinicaltrials.gov/large-docs/92/NCT03570892/SAP_001.pdf